CLINICAL TRIAL: NCT00642993
Title: A Multicenter, Randomized, Parallel-Group, Placebo-Controlled, Efficacy and Safety Trial to Evaluate the Effect of SCH 497079 on Weight in Obese and Overweight Subjects
Brief Title: Efficacy and Safety Trial to Evaluate the Effect of SCH 497079 on Weight in Obese and Overweight Participants (Study P05483)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05483; MK-7079-008 (Other: Merck protocol number)
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Overweight; Body Weight
MeSH Terms: conditions — Obesity; Overweight; Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCH 497079 (Experimental): SCH 497079, administered orally, once daily
  Interventions: Drug: SCH 497079
- Placebo (Placebo Comparator): Placebo capsules, administered orally, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCH 497079 — 100 mg capsule administered orally
  Arms: SCH 497079
Drug: Placebo — Placebo capsules matching SCH 497079 administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of SCH 497079 on weight in obese and overweight participants. The primary measure of effectiveness is the change in body weight during treatment. Additional measures include waist circumference and body mass index (BMI). In addition, the safety of SCH 497079 in obese and overweight participants will be evaluated. The primary hypothesis is that treatment with SCH 497079 will be more efficacious than that with placebo with respect to the primary efficacy variable.

DETAILED DESCRIPTION:
Following Screening, eligible participants will enroll in a Run-in Period. Participants who qualify for continuation in the study according to the entry criteria will be randomized to one of two treatment groups (SCH 497079 or placebo in a 2:1 ratio) with stratification according to gender.

Baseline measurements for the primary efficacy endpoint, as well as secondary endpoints will be evaluated at the Randomization Visit (Visit 3). Following randomization, participants will be treated for 12 weeks with double-blind study drug as adjunct to a 500 kcal deficit diet.

Participants will have scheduled visits after the Randomization Visit at 2 to 4 week intervals. Each participant will be encouraged to adhere to medication and dietary instructions.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age, of either sex, and of any race.
* Obese or overweight participants.

Exclusion Criteria:

* Participants who have a history of major eating disorders, gastrointestinal (GI) surgery, active serious cardiovascular, pulmonary, endocrine, neurologic, infectious, GI, hepatic, renal, hematologic, immunologic or psychiatric disease or diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2008-06-09 (Actual); Primary Completion 2009-01-30 (Actual); Study Completion 2009-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SCH 497079 | Placebo
Started | 267 | 134
Completed | 161 | 118
Not Completed | 106 | 16
Not completed — Adverse Event | 85 | 4
Not completed — Lost to Follow-up | 8 | 4
Not completed — Withdrew - reason unrelated to treatment | 11 | 3
Not completed — Protocol Violation | 1 | 4
Not completed — Did not meet protocol eligibility | 0 | 1
Not completed — Administrative | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCH 497079 | Placebo | Total
Number analyzed (Participants) | 267 | 134 | 401
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.2 (9.9) | 52.8 (10.4) | 53.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 93 | 279
  Male | 81 | 41 | 122

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Body Weight at Week 12
Description: Participant's body weight was measured in kilograms. For participants who discontinued during the study, last observation carried forward (LOCF) approach was applied to the analysis. any dropout before Week 12 was included in the analysis if the participant had a valid baseline and at least one post-baseline value.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population consisted of all participants who received randomized treatment assignment and had the baseline body weight measurement and at least one post-baseline body weight measurement.
Measure: Mean (Standard Error); unit: Kilogram
Arm/Group | SCH 497079 | Placebo
Number analyzed (Participants) | 255 | 130
Kilogram | -0.51 (0.19) | -0.92 (0.26)
Statistical Analysis 1: Comparison: SCH 497079 vs Placebo; Test type: Superiority or Other; p = 0.187, ANOVA; Mean and standard error are least squares means and corresponding standard errors based on an ANOVA model with main effects for treatment; Difference in means = 0.41, 95% CI 2-sided [-0.20 to 1.03]

2. Secondary Outcome: Percentage of Participants Demonstrating a Weight Loss ≥5% at Week 12
Description: For participants who discontinued during the study, LOCF approach was applied to the analysis. any dropout before Week 12 was included in the analysis if the participant had a valid baseline and at least one post-baseline value.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | SCH 497079 | Placebo
Number analyzed (Participants) | 255 | 130
Percentage of participants | 7.1 | 11.5
Statistical Analysis 1: Comparison: SCH 497079 vs Placebo; Test type: Superiority or Other; p = 0.140, Cochran-Mantel-Haenszel; The P-value is from the Cochran-Mantel-Haenszel Test adjusting for gender; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.28 to 1.20]

3. Secondary Outcome: Percentage of Participants Demonstrating a Weight Loss ≥10% at Week 12
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | SCH 497079 | Placebo
Number analyzed (Participants) | 255 | 130
Percentage of participants | 1.6 | 0.8
Statistical Analysis 1: Comparison: SCH 497079 vs Placebo; Test type: Superiority or Other; p = 0.515, Cochran-Mantel-Haenszel; The p-value is from the Cochran-Mantel-Haenszel Test adjusting for gender; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.24 to 9.93]

4. Secondary Outcome: Mean Change From Baseline in Waist Circumference at Week 12
Description: Participant's waist circumference was measured in centimeters. For participants who discontinued during the study, LOCF approach was applied to the analysis. any dropout before Week 12 was included in the analysis if the participant had a valid baseline and at least one post-baseline value.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Centimeters
Arm/Group | SCH 497079 | Placebo
Number analyzed (Participants) | 242 | 126
Centimeters | -1.22 (0.29) | -0.94 (0.39)
Statistical Analysis 1: Comparison: SCH 497079 vs Placebo; Test type: Superiority or Other; p = 0.543, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.20 to 0.63]

5. Secondary Outcome: Mean Change From Baseline in Body Mass Index (BMI) at Week 12
Description: For participants who discontinued during the study, LOCF approach was applied to the analysis. any dropout before Week 12 was included in the analysis if the participant had a valid baseline and at least one post-baseline value.
  Per protocol, participants were either obese (BMI ≥30 kg/m^2 and ≤40 kg/m^2) or overweight (BMI ≥27 kg/m^2 and <30 kg/m^2) at enrollment.
Time Frame: Baeline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | SCH 497079 | Placebo
Number analyzed (Participants) | 255 | 130
kg/m^2 | -0.18 (0.07) | -0.32 (0.09)
Statistical Analysis 1: Comparison: SCH 497079 vs Placebo; Test type: Superiority or Other; p = 0.231, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.09 to 0.35]

ADVERSE EVENTS:
Time Frame: Serious adverse events: Up to 16 weeks (including 30 days after the last dose of study drug); non-serious adverse events: up to 12 weeks
Arm/Group | SCH 497079 | Placebo
Serious Adverse Events (participants affected / at risk) | 5/267 | 1/134
Other Adverse Events (participants affected / at risk) | 142/267 | 26/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 497079 (N=267) | Placebo (N=134)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 497079 (N=267) | Placebo (N=134)
Nausea (Gastrointestinal disorders) | 35 (40) | 0 (0)
Nasopharyngitis (Infections and infestations) | 14 (14) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 18 (19) | 11 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Dysgeusia (Nervous system disorders) | 16 (16) | 0 (0)
Headache (Nervous system disorders) | 24 (25) | 1 (1)
Anxiety (Psychiatric disorders) | 18 (21) | 1 (1)
Insomnia (Psychiatric disorders) | 83 (91) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.